CLINICAL TRIAL: NCT04734938
Title: The Effect on Micronutrient Status of a Diet of 100% Huel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2003/4657
Record Dates: First submitted 2020-10-08; First posted 2021-02-02 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2020-10

CONDITIONS: Micronutrients
Keywords: Micronutrients

STUDY DESIGN:
Intervention Model Description: Open label crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual Diet (No Intervention): All volunteers will participate in this arm, continuing this habitual diet for 1 week
- 100% Huel (Experimental): All volunteers will participate in this arm of the study and consumer 100% Huel as their food for 4 weeks
  Interventions: Dietary Supplement: Huel Powder

INTERVENTIONS:
Dietary Supplement: Huel Powder — Huel is made of an ultra-fine blend of sustainable ingredients. Oats, rice, peas, coconut, flaxseed, and our unique mix of vitamins and nutrients to provide you a meal with all the carbohydrates, protein, essential fats, fibre, and all the 26 essential vitamins and minerals your body needs to thrive. Volunteers will consume only Huel as their food source for the final four weeks of the study.
  Arms: 100% Huel

SUMMARY:
This project will assess the effect of Huel Food replacement on the micronutrient status of healthy volunteers over a 4-week period.

To achieve this, 30 (non-smoking) generally healthy volunteers will be recruited to attend the study centre on three separate occasions. Volunteers will be asked to consume their normal diet for one week whilst recording what they eat. They will then be asked to only consume Huel Powder and water for 4 weeks.

DETAILED DESCRIPTION:
Study Protocol The effect on Micronutrient Status of a diet of 100% Huel

Aims of the study This project will assess the effect of Huel Powder on 30 generally healthy individuals over 4 weeks on the volunteer's micronutrient status. The aim is to identify any changes in the micronutrient status of volunteers in any of the 20 micronutrients to be monitored. Micronutrient status will be measured at the start of the study, after one week of their habitual diets and again after four weeks of consuming Huel powder as their single food source.

Huel Powder is a nutritionally complete powdered food that is high in protein and fibre, essential fats, carbohydrates, rich in phytonutrients and all 26 essential vitamins and minerals, with further information on Huel's website https://huel.com/pages/what-people-ask-about-huel.

Secondary measures of BMI, weight, waist and hip circumferences, and body composition will also be taken to observe any changes over the study period.

All researchers will be trained in GCP and phlebotomy. Potential volunteers will sent a health and activity questionnaire to assess their energy consumption and expenditure. This can be discussed over a Zoom call (or similar platform) if required. This will be used to screen the volunteers to see if they are suitable for the study. The energy intake information will also be verified from the first week of the study when they are consuming their habitual diet and completing their food diaries on my fitness pal. The energy requirements will inform the researcher how much Huel the volunteers will require over the course of the four weeks.

The volunteers will come to the study centre at Newcastle on three separate occasions. The first, at the start of the study they can have any further questions answered and if they are happy to take part in the study, they will be asked to complete a written consent form. They will also have their height, weight, body composition, waist and hip circumferences, measured as well as giving a blood sample (30ml) for micronutrient analysis. The second visit, at the end of the first week, will also measure the weight, body composition, waist circumference and take a blood sample. The final visit will be at the end of the study taking weight, body composition, waist circumference and a blood sample for micronutrient analysis.

The micronutrients and blood markers to be measure are listed below.

Markers to be tested; Haemoglobin Sodium Calcium HbA1c Cholesterol status Iron status Vitamin A Vitamin D Vitamin E Vitamin C Folate Vitamin B12 Choline Magnesium Potassium Zinc Copper Manganese Selenium Iodine (TSH)

Analysis Plan Although this trial is a pilot study, changes in BMI, weight, body composition, waist circumference, and micronutrient/blood marker will be compared between 0 and 1 week, as well as 1 week and 5 weeks, will be assessed. A one-way ANOVA will be used to assess differences for individual volunteers.

Test conditions Each volunteer will be asked to continue to consume their habitual diet for the first week and record their food intake in food diary app, myfitnesspal. At the end of the first week volunteers will be asked to consume only the Huel Powder provided and water. Volunteers will be asked not to consume any other food or drinks during these four weeks but still record their Huel intake in myfitnesspa.

* 100% Huel - Only a diet comprising of Huel powder must be consumed for the last four weeks of the trial. No other snacks/food are permitted.
* Energy intake - Daily calorie requirements varies from person to person and is determined by weight, height, gender, age and activity levels. The researchers will help estimate individual calorie requirements. Once you have your calorie requirements, manipulate your Huel serving sizes to reflect daily calorie intake.
* Huel products - Only Huel powder - as well as Huel Flavour Boosts, if desired - must be consumed as part of this study. Huel Granola or Huel Bars cannot be consumed during this study.
* Fluid intake - Only plain water, herbal tea (excluding citrus teas), black tea or coffee must be drunk. No additions must be made to fluid, i.e. no additional sugar, sweeteners, milk or honey are permitted during the length of the study.
* Alcohol intake - No alcohol must be consumed during the study.
* Exercise/Activity- Participants are able to continue with normal exercise and activity during the study.

Volunteers Thirty generally healthy volunteers, males and nonpregnant, nonlactating females aged over 18 years will be recruited for the study. Volunteers will be recruited by posters and word of mouth from Newcastle University staff and their associates.

Anonymity

Volunteers will be assigned a 'Participant Identification Number', which volunteers will use to complete questionnaires and researcher will use to label volunteers blood samples. Ony one documents will contain volunteers names and Participant Identification Number, and this will be destroyed after the final volunteer has completed the study or once the study has been concluded, which ever occurs first. Consent forms will not contain Participant Identification Numbers and will be kept for 12 months after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* generally health (includes not having been diagnosed with any eating disorders and not receiving regular medication other than contraceptives or statins)
* 18 years or older,
* non-pregnant,
* non-lactating
* non-smoking,
* no known food allergies.

Exclusion Criteria:

*taking medication for long term illnesses such as high blood pressure, heart disease, or medication that affects liver or kidney function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Change in level of calcium, cholesterol status, haemoglobin, magnesium, sodium, potassium in blood | week 0 and week 1
  Change in the level of alcium, cholesterol status, haemoglobin, magnesium, sodium, potassium in blood (mmol/l)
Change in level of calcium, cholesterol status, haemoglobin, magnesium, sodium, potassium in blood | week 1 and week 5
  Change in the level of calcium, cholesterol status, haemoglobin, magnesium, sodium, potassium in blood (mmol/l)
Change in level of HbA1c in blood | week 0 and week 1
  Change in the level of HbA1c in blood (mmol/mol)
Change in level of HbA1c in blood | week 1 and week 5
  Change in the level of HbA1c in blood (mmol/mol)
Change in level of choline, copper, Iron status, selenium, Vitamin A, Vitamin C, Vitamin E, Vitamin D and Zinc | week 0 and week 1
  Change in the level of choline, copper, Iron status, selenium, Vitamin A, Vitamin C, Vitamin E, Vitamin D and Zinc in blood (micro mol/l)
Change in level of choline, copper, Iron status, selenium, Vitamin A, Vitamin C, Vitamin E, Vitamin D and Zinc | week 1 and week 5
  Change in the level of choline, copper, Iron status, selenium, Vitamin A, Vitamin C, Vitamin E, Vitamin D and Zinc in blood (micro mol/l)
Change in level of manganese and Folate | week 0 and week 1
  Change in the level of manganese and Folate in blood (nmol/l)
Change in level of manganese and Folate | week 1 and week 5
  Change in the level of manganese and Folate in blood (nmol/l)
Change in level of Vitamin B12 | week 0 and week 1
  Change in the level of Vitamin B12 in blood (pmol/l)
Change in level of Vitamin B12 | week 1 and week 5
  Change in the level of Vitamin B12 in blood (pmol/l)
Change in level of Thyroid Stimulating Hormone (TSH) | week 0 and week 1
  Change in the level of THS in blood (mU/l)
Change in level of Thyroid Stimulating Hormone (TSH) | week 1 and week 5
  Change in the level of THS in blood (mU/l)

SECONDARY OUTCOMES:
Change in BMI | Week 0 and week 1
  change in BMI (kg/m2)
Change in BMI | week 1 and week 5
  change in BMI (kg/m2)
Change in Weight | Week 0 and week 1
  change in weight (kg)
Change in Weight | week 1 and week 5
  change in weight (kg)
Change in hip to waist ratio | Week 0 and week 1
  change in hip to waist ratio
Change in hip to waist ratio | week 1 and week 5
  change in hip to waist ratio
Change in body composition of fat | week 0 and week1
  change in body composition of fat (%) as measured by impedance
Change in body composition of fat | week 1 and week 5
  change in body composition of fat (%) as measured by impedance

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Pearson, PhD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle University, Newcastle, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No